CLINICAL TRIAL: NCT04389125
Title: 12 Weeks, Randomized, Double-blind, Placebo-controlled Human Trial to Evaluate the Efficacy and Safety of Angelica Gigas Nakai and Allium Cepa L.Extract Mixtures on the Improvement of Blood Flow
Brief Title: Efficacy and Safety of Angelica Gigas Nakai and Allium Cepa L.Extract Mixtures on the Improvement of Blood Flow
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chonbuk National University Hospital (Other)
Responsible Party: Principal Investigator, Soo-Wan Chae, Principal Investigator, Clinical Trial Center for Functional Foods, Chonbuk National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: HJ-BF-AAM
Record Dates: First submitted 2020-04-29; First posted 2020-05-15 (Actual); Last update posted 2020-05-15 (Actual); Status verified 2020-05

CONDITIONS: Blood Flow

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Improvement of Blood Flow group (Experimental): One packet once a day, after breakfast (1.5 g/day, 1.5 g/day as an Angelica Gigas Nakai and Allium Cepa L.Extract Mixtures)
  Interventions: Dietary Supplement: Angelica Gigas Nakai and Allium Cepa L.Extract Mixtures
- Placebo group (Placebo Comparator): One packet once a day, after breakfast (1.5 g/day)
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Angelica Gigas Nakai and Allium Cepa L.Extract Mixtures — One packet once a day, after breakfast, for 12 week
  Arms: Improvement of Blood Flow group
Dietary Supplement: Placebo — Placebo for 12 week
  Arms: Placebo group

SUMMARY:
This study was conducted to investigate the effects of daily supplementation of Angelica Gigas Nakai and Allium Cepa L.Extract Mixtures on the Improvement of Blood Flow.

DETAILED DESCRIPTION:
This study was a 12-week, randomized, double-blind, placebo-controlled human trial. 80 subjects were randomly divided into Angelica Gigas Nakai and Allium Cepa L.Extract Mixtures group and a placebo group. It is to evaluate the changes in the displayed evaluation items when taking Angelica Gigas Nakai and Allium Cepa L.Extract Mixtures once a day, in comparison with taking a placebo.

ELIGIBILITY:
Inclusion Criteria:

* Participants who meet three or more items
* Smoker
* Total cholesterol 180~239 mg/dL before a meal
* LDL cholesterol 130~159 mg/dL before a meal
* Glucose 100~125 mg/dL before a meal
* systolic blood pressure(SBP) is 120~140 mmHg
* Body mass index(BMI) is 23~30 kg/m^2
* Waist/Hip ratio(WHR) is 0.9 over for man, 0.85 over for a woman

Exclusion Criteria:

* Participants with marked impairment of platelet function and platelet coagulation
* Participants who have anticoagulation within 4 weeks before the screening test
* Participants with a clinically significant acute or chronic cardiovascular system, endocrine system, immune system, respiratory system, liver biliary system, kidney and urinary system, neuropsychiatry system, musculoskeletal system, Inflammation, blood tumor, gastric disease, etc.
* Participants with BMI(Body mass index) less than 18.5 kg/m^2 or more than 35 kg/m^2 at the screening test
* Participants who take medicine or healthy functional foods for platelet function, blood circulation improvement, and hyperlipidemia within 4 weeks before the screening test
* Participants receiving antipsychotic medication within 3 months prior to the screening test
* Participants suspected of alcoholism(21 unit/week) or substance abuse
* Participants who have participated in other clinical trials within 3 months prior to the screening test
* Participants who show the following relevant results in a Laboratory test º Aspartate Transaminase(AST), Alanine Transaminase(ALT) > Reference range 3 times upper limit º Serum Creatinine > 2.0 mg/dl
* Women who are pregnant or breastfeeding
* Women who may become pregnant and have not used appropriate contraceptives
* Participants who the principal investigator judged inappropriate for the participant in this study because of a laboratory test result, etc

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2020-01-30 (Actual); Primary Completion 2021-04-30 (Estimated); Study Completion 2021-05-30 (Estimated)

PRIMARY OUTCOMES:
Changes of Platelet function assay(PFA) | Baseline, 12 week
  The concentration of Platelet function assay(PFA) was assessed before and after the intervention
Changes of blood viscosity | Baseline, 12 week
  The concentration of blood viscosity was assessed before and after the intervention

SECONDARY OUTCOMES:
Changes of systolic blood pressure(SBP), diastolic blood pressure(DBP), Pulse | screening, 0 week, 6 week, 12 week
  systolic blood pressure(SBP), diastolic blood pressure(DBP), Pulse were measured in study screening, visit 1(0 week), visit 2(6 weeks) and visit 3(12 weeks).
Changes of blood coagulation-related indices | Baseline, 12 week
  Blood coagulation-related indices(e.g. Plasminogen activator inhibitor-1, Serotonin, Thromboxane B2, activated partial thromboplastin time) were measured in study visit 1(0 week) and visit 3(12 weeks).
Changes of indicator of lipid metabolism | Baseline, 12 week
  Lipid metabolism(e.g. Total cholesterol, Triglyceride, Low Density Lipoprotein-cholesterol, High Density Lipoprotein-cholesterol, Non High Density Lipoprotein-cholesterol) was measured in study visit 1(0 week) and visit 3(12 weeks).
Changes of atherosclerosis index | Baseline, 12 week
  Atherosclerosis index(e.g. Total cholesterol/High Density Lipoprotein-cholesterol, Low Density Lipoprotein-cholesterol/High Density Lipoprotein-cholesterol, Triglyceride/High Density Lipoprotein-cholesterol, (Total cholesterol-High Density Lipoprotein-cholesterol)/High Density Lipoprotein-cholesterol) was measured in study visit 1(0 week) and visit 3(12 weeks).

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Trial Center for Functional Foods Chonbuk National University Hospital, Jeonju, Jeollabuk-do, South Korea